CLINICAL TRIAL: NCT01293604
Title: The Influence of Daily Intake of Whole Grain Barley or Oats on Biomarkers of Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Collaborators: Kellogg Company (Industry)
Responsible Party: Janet A. Novotny, USDA
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HS34
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Barley; Oats; Whole grains; Cardiovascular disease; adults not taking lipid-lowering or glucoregulatory medications.
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whole Grain Barley Diet (Experimental): A controlled diet containing at least 4 daily servings of whole grain barley.
  Interventions: Other: Daily ingestion of whole grain barley and oats
- Whole Grain Oats Diet (Active Comparator): A diet containing at least 4 servings of whole grain oats.
  Interventions: Other: Daily ingestion of whole grain barley and oats
- Low Whole Grain Diet (Other): A control diet containing 0.7 daily servings of whole grain.
  Interventions: Other: Daily ingestion of whole grain barley and oats

INTERVENTIONS:
Other: Daily ingestion of whole grain barley and oats — Subjects will be randomly assigned to one of three treatments: 1) a control diet containing 0.7 daily servings of whole grain, 2) a diet containing at least 4 daily servings of whole grain barley or 3) a diet containing at least 4 servings of whole grain oats. After 6 weeks, risk factors of cardiovascular disease will be assessed after a 12 hr fast. During the seventh week, risk factors of cardiovascular disease will be assessed in the postprandial state.

SUMMARY:
The objectives of this study are the following: 1) to determine the effect of daily consumption of whole grain barley for six week on risk factors of cardiovascular disease compared to a diet low in whole grains, and 2) to compare the effects of daily consumption of whole grain barley to those of whole grain oats for six weeks to determine if the response to these two grains is different.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 25-70 years
* Body mass index (BMI) ≥ 19 and ≤ 38
* Willingness and ability to make scheduled appointments at clinical site as required by study protocol

Exclusion Criteria:

* Do not regularly consume breakfast or dislike cereal for breakfast
* Known (self-reported) allergy or adverse reaction to grains (e.g., wheat, gluten, barley)
* Presence of kidney disease, liver disease, gout, untreated or unstable hypothyroidism, untreated or unstable hyperthyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* Fasting triglycerides > 300 mg/dL
* Fasting glucose > 126 mg/dL
* Use of cholesterol lowering medication
* Blood pressure > 180/100 or hypertension treated with calcium channel blockers, direct acting vasodilators, or beta blockers
* History of bariatric or certain other surgeries related to weight control
* History of major surgery within 3 months of enrollment
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* Antibiotic use during the intervention or for 3 months prior to the intervention period
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 6 months
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Meal Tolerance Assessment | 7 hours
  Subjects will provide a baseline blood sample at 15 minutes and 5 minutes prior to consuming a test meal. Subjects will then consume a high fat breakfast of foods such as eggs, buttered English muffins, and donuts. Blood samples will be collected 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 360, and 420 min following ingestion of the test meal. Measurements will be made for serum triglyceride area under the curve, serum cholesterol, insulin, glucose, and plasma apo B48.
Biomarkers of cardiovascular risk | After a 12 hour fast
  Fibrinogen, factor VII, blood pressure, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, Lp(a), and lipoprotein size.
Biomarkers of oxidative stress | After 6 weeks of feeding
  Nitrites and nitrates, malondialdehyde, lipid hydroperoxides, ox-LDL, resistance of LDL to Cu2+-induced oxidation, FRAP, glutathione, glutathione-S-transferase, super oxide dismutase, PON-1, betaine, homocysteine, total thiols, urinary isoprostanes.
Biomarkers of inflammation | After 6 weeks of controlled feeding
  C-reactive protein (CRP), IL-6, IL-8, IL-10, IL-18, TNFα, matrix metalloproteinases (MMP-2, MMP-9), e-Selectin, ICAM, VCAM
Biomarkers of glucoregulatory control | After 6 weeks of feeding
  Glycated apolipoprotein B, hemoglobin A1c, fructosamine, insulin, glucose, leptin, adiponectin

SECONDARY OUTCOMES:
Genotype testing | After 6 weeks of controlled feeding
  Blood will be used to test for genetic traits that may influence nutrient metabolism and also traits reflecting the mechanisms that may be influenced by the intervention.
Microarray and targeted gene expression testing | After 6 weeks of controlled feeding
  Blood samples will be used to test how the intervention affects gene expression. Global gene expression will be performed for a complete survey of the RNA response to the intervention. Targeted gene expression will be performed to confirm the findings of the global gene expression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Janet A Novotny, PhD, Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States